CLINICAL TRIAL: NCT02222753
Title: Therapeutic Effect and Prognosis Predication Related Immunocyte Subgroup and Immunologic Factors Screeing for Colorectal Cancer
Brief Title: Immunological Markers Screening for Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: State Key Laboratory of Cancer Biology (Network)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other); Air Force Military Medical University, China (Other); Second Military Medical University (Other); China-Japan Friendship Hospital (Other); Chinese Academy of Medical Sciences (Other); Peking University Cancer Hospital & Institute (Other); Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dake Chu, Dr., State Key Laboratory of Cancer Biology
Other Study IDs: 2014AA020801
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blood specimens
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Colorectal cancer incidence is increasing at an alarming rate in China. Recent reports concluded aberrant immunological function was associated with colorectal cancer outcome, however, the influence of immunocyte subgroup and immunologic factors on cancer outcome in colorectal cancer survivors is largely unknown.The investigators will explore the impact of immunocyte subgroup and immunologic factors on colorectal cancer disease-specific, disease-free and overall survival. The investigators will recruit approximately 5,000 patients as a prospective study cohort. During follow up, the investigators will explore the association of these factors with outcome of patients. The investigators believe that this project will improve the understanding of the impact of immunocyte subgroup and immunologic factors on colorectal cancer outcome.

ELIGIBILITY:
Inclusion Criteria:

Patient must have a histologically proven adenocarcinoma of colon or rectum cancer.

* Patients must have a performance status of 0,1, or 2 by the Southwest Oncology Group criteria.
* Patients must have recovered from any effects of surgery.
* Evaluable disease must be present outside radiation field. At least 3 weeks must have elapsed after discontinuation of radiation therapy.
* Patients must provide a signed consent to participate in the study.
* Patients must complete all questionnaires.

Exclusion Criteria:

Patients with a proven history of peptic ulcer disease or gastroesophageal reflux.

* History of other malignancy, except for cancers that have been treated with a curative intent and patient is without evidence of active disease.
* Unresolved bacterial infection requiring treatment with antibiotics.
* Pregnant or lactating women may not participate in the study.
* Patients known to have HIV-1 virus infection because of the undetermined effect of this chemotherapy regimen in patients with HIV-1 and the potential for serious interaction with anti-HIV medications.
* Gilbert's disease.
* Other serious concurrent infection
* Clinically significant cardiac disease not well controlled with medication (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias) or myocardial infarction within the last 12 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Disease-specific survival | 5 years
  Disease-specific survival is defined as the time elapsed from surgery to death due to CRC. Concretely, the cause of death obtained in the follow up was classified according to ICD-10 conventions. Disease-specific deaths included those with an underlying cause attributed to ICD-10 codes C18.0-C20.0 or C26.0.

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival is defined as the time elapsed from surgery to the date of death from any cause.

OTHER OUTCOMES:
Disease-free survival | 5 years
  Disease-free survival is defined as the time elapsed from surgery to the first occurrence of any of the following events: recurrence of colorectal cancer; colorectal cancer distant metastasis; development of second non-colorectal malignancy excluding basal cell carcinomas of the skin and carcinoma in situ of the cervix; or death from any cause without documentation of a cancer-related event.

CONTACTS AND LOCATIONS:
Overall Officials: Long Cui, M.D., Study Chair — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China